CLINICAL TRIAL: NCT02467868
Title: Multicenter, Double-Blind, Randomized, Comparative Efficacy and Safety Study of MYL-1401H and European Sourced Neulasta® in Stage II/III Breast Cancer Patients Receiving Neoadjuvant or Adjuvant Chemotherapy
Brief Title: Efficacy and Safety Study With MYL-1401H and Neulasta
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: Mylan GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MYL-1401H-3001; 2014-002324-27 (EudraCT Number)
Record Dates: First submitted 2015-06-08; First posted 2015-06-10 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Breast Neoplasms; Chemotherapy-Induced Febrile Neutropenia
Keywords: Pegfilgrastim; Granulocyte Colony Stimulating Factor (G-CSF); Breast Cancer; Neutropenia
MeSH Terms: conditions — Breast Neoplasms; Chemotherapy-Induced Febrile Neutropenia; Neutropenia | interventions — MYL-1401H; pegfilgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MYL-1401H (Experimental): MYL-1401H
  Interventions: Biological: MYL-1401H
- Neulasta (Active Comparator): Neulasta
  Interventions: Biological: Neulasta

INTERVENTIONS:
Biological: MYL-1401H — During each chemotherapy cycle MYL-1401H (6 mg) is administered s.c. 24 hours after chemotherapy.
  Other Names: Pegfilgrastim; Recombinant human granulocyte colony-stimulating factor (G-CSF)
  Arms: MYL-1401H
Biological: Neulasta — During each chemotherapy cycle Neulasta (6 mg) is administered s.c. 24 hours after chemotherapy.
  Other Names: Pegfilgrastim; Recombinant human granulocyte colony-stimulating factor (G-CSF)
  Arms: Neulasta

SUMMARY:
This is a Multicenter, Double-Blind, Randomized, Comparative Efficacy and Safety Study of MYL-1401H and Neulasta (Pegfilgrastim) in Stage II/III Breast Cancer Patients Receiving Neoadjuvant or Adjuvant Chemotherapy.

DETAILED DESCRIPTION:
After successful screening, eligible patients will be randomly allocated to one of the two study arms, either receiving MYL-1401H or Neulasta.

Randomization is 2:1 to MYL-1401H or Neulasta, respectively.

Subjects will receive first of six cycles of background therapy (Docetaxel, Doxorubicin, Cyclophosphamide [TAC]) on day 1. Treatment with study drug (either MYL-1401H or Neulasta) is scheduled on Day 2 of each cycle, at least 24 hours after chemotherapy administration.

Duration of each cycle is 3 weeks.

Follow-up visit is scheduled 24 weeks after the first administration of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent.
* Patients ≥18 years.
* Women of child-bearing potential must agree to use effective methods of birth control during the treatment period from the first dose of study drug until 6 months following the last dose of study drug.
* Newly diagnosed, pathologically confirmed breast cancer.
* Stage II or III breast cancer with adequate staging workup and adequate surgery if receiving adjuvant therapy.
* Patients planned/eligible to receive neoadjuvant or adjuvant treatment with (Docetaxel, Doxorubicin, Cyclophosphamide [TAC]) for their breast cancer.
* Cancer Chemotherapy and Radiotherapy naïve.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Absolute neutrophil count ≥ 1.5 × 109/L ; Platelet count ≥ 100 × 109/L ;
* Hemoglobin > 10 g/dL without blood transfusions or cytokine support during the two weeks previous to the hemoglobin level.
* Adequate cardiac function (including left ventricular ejection fraction ≥ 50% as assessed by echocardiography) within 4 weeks prior to start of chemotherapy.
* Adequate renal function, i.e., creatinine < 1.5 × upper limit of normal (ULN).

Other protocol specific inclusion/exclusion criteria may apply

Exclusion Criteria:

* Participation in a clinical trial in which they received an investigational drug within 28 days before randomization.
* Previous exposure to filgrastim, pegfilgrastim, lenograstim, lipegfilgrastim, or other filgrastim forms on the market or in clinical development.
* Received blood transfusions or erythroid growth factors within 2 weeks prior to first dose of chemotherapy.
* Known hypersensitivity to any drugs or excipients that patients will be receiving during the study.
* Known hypersensitivity to E. coli-derived products.
* Known fructose intolerance (related with sorbitol excipient).
* Underlying neuropathy of grade 2 or higher.
* Active infectious disease or any other medical condition which might put the patient at significant risk to tolerate 6 courses of TAC chemotherapy (e.g., recent myocardial infarction).
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 × Upper limit of normal (ULN), ALT and/or AST > 1.5 × ULN with alkaline phosphatase (ALP) > 2.5 × ULN; any bilirubin > ULN.
* Treatment with systemically active antibiotics within 5 days before first dose of chemotherapy.
* Patients under treatment with lithium.
* Chronic use of oral corticosteroids.
* Splenomegaly of unknown origin by physical examination and/or computerized tomography scan or ultrasound and any condition which can cause splenomegaly, e.g., thalassemia, glandular fever, hemolytic anemias, and malaria.
* Myeloproliferative or myelodysplastic disorders, sickle cell disorders, and any illness or condition that in the opinion of the investigator may affect the safety of the patient or the evaluation of any study endpoint.
* Increase potential risk of Adult Respiratory Distress Syndrome.
* Pregnant or nursing women.
* Patients known to be seropositive for human immunodeficiency virus (HIV), or who have had an acquired immunodeficiency syndrome (AIDS) defining illness or a known immunodeficiency disorder.
* A known active abuse of drugs or alcohol should preclude patient participation and evaluation in the study.
* Any known psychiatric conditions.
* Any disease or physical condition that may not allow for the adequate performance of study assessments, such as lack of access to patient's domiciliary, and distance of patient's domiciliary from clinic site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Mean Duration of Severe Neutropenia (DSN), defined as consecutive days with absolute neutrophil count (ANC) < 0.5 × 109/L | Cycle 1 of chemotherapy (approx 21 days)

SECONDARY OUTCOMES:
The rate of febrile neutropenia (FN) | Week 24 (End of the study)

OTHER OUTCOMES:
Incidence, nature, and severity of adverse events (AEs) | Week 24
  Rate of FN listed by cycles and across cycles
Presence of antibodies against MYL-1401H and Pegfilgrastim | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus Rojkjaer, MD, Study Chair — Mylan GmbH
Locations (36):
- Bulgaria (7):
  - Mylan Investigational Site 3502, Plovdiv
  - Mylan Investigational Site 3506, Plovdiv
  - Mylan Investigational Site 3507, Plovdiv
  - Mylan Investigational Site 3503, Sofia
  - Mylan Investigational Site 3505, Sofia
  - Mylan Investigational Site 3504, Varna
  - Mylan Investigational SIte 3501, Veliko Tarnovo
- Georgia (7):
  - Mylan Investigational Site 9901, Tbilisi
  - Mylan Investigational Site 9902, Tbilisi
  - Mylan Investigational Site 9903, Tbilisi
  - Mylan Investigational Site 9904, Tbilisi
  - Mylan Investigational Site 9905, Tbilisi
  - Mylan Investigational Site 9906, Tbilisi
  - Mylan Investigational Site 9907, Tbilisi
- Mylan Investigational site 4905, Bonn, Germany
- Hungary (8):
  - Mylan Investigational Site 3604, Budapest
  - Mylan Investigational SIte 3606, Budapest
  - Mylan Investigational Site 3607, Budapest
  - Mylan Investigational Site 3609, Debrecen
  - Mylan Investigational Site 3601, Gyula
  - Mylan Investigational SIte 3605, Nyíregyháza
  - Mylan Investigational Site 3603, Szombathely
  - Mylan Investigational Site 3602, Zalaegerszeg
- Poland (3):
  - Mylan Investigational site 4802, Bydgoszcz
  - Mylan Investigational Site 4805, Kościerzyna
  - Mylan Investigational SIte 4804, Krakow
- Ukraine (10):
  - Mylan Investigational SIte 3804, Chernivtsi
  - Mylan Investigational site 3801, Dniepropetrovsk
  - Mylan Investigational Site 3805, Dniepropetrovsk
  - Mylan Investigational Site 3808, Kharkiv
  - Mylan Investigational Site 3810, Kyiv
  - Mylan Investigatational Site 3802, Lutsk
  - Mylan Investigational SIte 3807, Lviv
  - Mylan Investigational SIte 3803, Odesa
  - Mylan Investigational Site 3809, Sumy
  - Mylan Investigational Site 3806, Uzhhorod

REFERENCES:
- [Derived] Waller CF, Ranganna GM, Pennella EJ, Blakeley C, Bronchud MH, Mattano LA Jr, Berzoy O, Voitko N, Shparyk Y, Lytvyn I, Rusyn A, Popov V, Lang I, Beckmann K, Sharma R, Baczkowski M, Kothekar M, Barve A. Randomized phase 3 efficacy and safety trial of proposed pegfilgrastim biosimilar MYL-1401H in the prophylactic treatment of chemotherapy-induced neutropenia. Ann Hematol. 2019 May;98(5):1217-1224. doi: 10.1007/s00277-019-03639-5. Epub 2019 Mar 1. PMID 30824956